CLINICAL TRIAL: NCT00183846
Title: Phase I Study of Irinotecan Administered as a Continuous Infusion and Radiation Therapy for Upper Gastrointestinal Cancers
Brief Title: Study of Irinotecan Administered as a Continuous Infusion and Radiation Therapy for Upper Gastrointestinal Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0C-00-8
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Cancer; Gastric Cancer; Duodenum Cancer; Bile Duct Cancer
Keywords: pancreas; stomach; common bile duct cancer; ampulla of Vater cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Duodenal Neoplasms; Bile Duct Neoplasms | interventions — Irinotecan; Radiotherapy

INTERVENTIONS:
Drug: irinotecan
Procedure: radiation therapy

SUMMARY:
This study is for people with advanced cancer of the digestive tract and cancer that cannot be completely removed by surgery. Radiation therapy is commonly used in the treatment of these types of cancer in combination with a chemotherapy drug, called 5-fluorouracil (5-FU). In this study, doctors will administer the standard dose of radiation therapy in combination with an investigational chemotherapy drug, called irinotecan. Irinotecan can decrease the size of tumors and also appears to increase the effectiveness of radiation. The purpose of this study is to determine the highest dose of irinotecan that can be given safely in combination with radiation therapy, and to determine the side effects when these two treatments are given together. Irinotecan is approved by the Food and Drug Administration (FDA) for the treatment of colon cancer, but is not approved for cancers of the digestive tract. However, the FDA is allowing its use in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed neoplasm of the upper gastrointestinal tract (pancreas, stomach, duodenum, common bile duct, ampulla of Vater) or metastatic tumor to the upper abdomen.
* Eligible patients include patients with locally advanced unresectable tumors, positive surgical margins, local recurrence and resected stage II-III pancreatic, gastric, duodenum, bile duct or ampulla of Vater carcinoma.
* Performance status SWOG 0-2
* Fully recovered from prior surgery or chemotherapy (greater than or equal to 4 weeks). Patients previously treated with 5-FU or gemcitabine may start therapy 2 weeks after the last dose of 5-FU or gemcitabine.
* Absolute granulocyte count (AGC) > 1500; platelets > 100,000; serum creatinine < 2.0 mg/dl; total bilirubin < 2.0 mg/dl; AST or ALT and alkaline phosphatase < 3 times the upper limit of normal.
* Prior chemotherapy is allowed.

Exclusion Criteria:

* Prior radiation therapy to the upper abdomen
* Tumors of the gastroesophageal junction.
* Other medical, psychological or social circumstances that, in the opinion of the investigator, would prevent participation in the clinical trial
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2000-12; Primary Completion 2007-10 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of irinotecan when administered as a 5-day continuous infusion with concomitant radiation therapy in patients with upper gastrointestinal tumors (pancreas, stomach, duodenum, and common bile duct)

SECONDARY OUTCOMES:
To describe the toxicity profile observed with this combination
To obtain preliminary information related to the efficacy of this combination

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — U.S.C./Norris Comprehensive Cancer Center
Locations (1):
- U.S.C./Norris Cancer Center, Los Angeles, California, United States